CLINICAL TRIAL: NCT04049019
Title: Biomarkers in Urine for Children With Monosymptomatic Nocturnal Enuresis and Nocturnal Polyuria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Biomarkers in MNE
Record Dates: First submitted 2019-08-01; First posted 2019-08-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Nocturnal Enuresis
MeSH Terms: conditions — Nocturnal Enuresis | interventions — Urine Specimen Collection

STUDY DESIGN:
Intervention Model Description: 10 boys with nocturnal enuresis and 10 healthy boys will be included for urine collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urine collection, children with nocturnal enuresis (Experimental): The child ́s weight and height will be registered. The children's urine will be tested for infection with a dipstick urinalysis.
  The child will be asked to perform home recordings for seven days consisting of measurements of diaper weight and first morning voided volume and a two-day frequency-volume chart.
  Interventions: Diagnostic Test: Urine collection through a collecting device (Uridome®) for maximum 1 week
- Urine collection, healthy children (Active Comparator): The child ́s weight and height will be registered. The children's urine will be tested for infection with a dipstick urinalysis.
  Interventions: Diagnostic Test: Urine collection

INTERVENTIONS:
Diagnostic Test: Urine collection through a collecting device (Uridome®) for maximum 1 week — The child will collect:
  * Urine at bedtime before a wet and a dry night.
  * Urine during a wet night through a collecting device.
  * First morning voided volume following both a wet and a dry night.
  Arms: Urine collection, children with nocturnal enuresis
Diagnostic Test: Urine collection — The child will collect:
  * Urine at bedtime.
  * First morning voided volume
  Arms: Urine collection, healthy children

SUMMARY:
The aim of the study is to identify protein markers in relation to the enuresis related nocturnal polyuria by using mass spectrometry on nocturnal urine samples. A biomarker for nocturnal polyuria would simplify an important part of the clinical characterization of enuresis patients.

DETAILED DESCRIPTION:
Involuntary voiding during sleep, nocturnal enuresis (NE), affects 7-10 % of all 7-year-olds, and 0.5-2 % of young adults. Night-time polyuria is one of the main pathogenic mechanisms. Today, the only method to diagnose nocturnal polyuria is home recordings involving diaper weight and registrations of first morning voids, which is very time-consuming. By using mass spectrometry (proteomics and metabolomics) on nocturnal urine samples from children with NE, the investigators aim to identify protein markers in relation to nocturnal polyuria. The perspective is to simplify an important part of the clinical characterization of NE patients.

This hypothesis-generating pilot project will be performed on 10 boys with NE. The children will have to collect:

* Urine at bedtime on a wet and a dry night.
* Urine during a wet night through a collecting device (non-invasive).
* First morning voided volume following both a wet and a dry night.

Furthermore, we will include 10 children without NE, who will collect urine during a dry night (first morning voided volume).

Endpoints are any biomarkers in urine found to be associated with nocturnal polyuria.

The proteomics and metabolomics methodologies are available at the proteomics core facility of Research Unit for Molecular Medicine, Dept. of Clinical Medicine, Aarhus University Hospital.

Based on the analytical uncertainty of the protein analysis methods, 10 samples are sufficient for detecting down to two-fold alterations in protein levels (p<0.05). By using state of the art mass spectrometry, the difference in any protein level between 1) the total urine amount on a wet and a dry night, and 2) first morning voided volume on a wet and a dry night, will be evaluated. Furthermore, difference in urine composition between children with NE and healthy children will be evaluated. Student's t-test with significance level at p<0.05 will be used.The amount of proteins in each urine sample will be correlated to the total amount of proteins in the respective sample.

ELIGIBILITY:
Inclusion Criteria:

* Monosymptomatic nocturnal enuresis with at least one dry night per week.
* Nocturnal polyuria defined as nocturnal urine production on wet nights greater than 130 % of expected bladder capacity for age.
* Normal bladder capacity defined as maximum voided volume excluding first morning voided volume bigger than expected bladder capacity for age.

Exclusion Criteria:

* Recurrent urinary tract infections.
* Anamnestic, clinical or laboratory findings that can be related to diseases or conditions that might affect the parameters investigated.
* Neurological and/or known clinically significant anatomical abnormalities of the urinary tract.
* Former operations in the urinary tract.
* Ongoing medication that may interfere with the parameters tested.

If the child is receiving treatment for nocturnal enuresis (desmopressin, alarm or anticholinergics), the treatment has to be paused 1 week before urine collection.

Furthermore, we will include 10 children without nocturnal enuresis and otherwise healthy.

Ages: 6 Years to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Proteins. | Up to 1 week.
  By using mass spectrometry (proteomics). For all children, any proteins related to nocturnal polyuria will be detected.
Metabolites. | Up to 1 week.
  By targeted mass spectrometry.

SECONDARY OUTCOMES:
Total urine volume in each sample. | Up to 1 week.
  A urine volume for the "dry night" (first morning voided volume) and "wet night" (nighttime urine production + first morning voided volume) will be calculated.
Concentration of creatinine in the urine samples. | Up to 1 week.
  A level for the "dry night" and "wet night" will be calculated.
Osmolality in the urine samples. | Up to 1 week.
  By freezing-point depression. A level for the "dry night" and "wet night" will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Søren Rittig, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Paediatrics and Adolescent Medicine, Aarhus University Hospital, Aarhus, Jylland, Denmark

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] von Gontard A, Heron J, Joinson C. Family history of nocturnal enuresis and urinary incontinence: results from a large epidemiological study. J Urol. 2011 Jun;185(6):2303-6. doi: 10.1016/j.juro.2011.02.040. Epub 2011 Apr 21. PMID 21511300
- [Background] Butler RJ, Heron J. The prevalence of infrequent bedwetting and nocturnal enuresis in childhood. A large British cohort. Scand J Urol Nephrol. 2008;42(3):257-64. doi: 10.1080/00365590701748054. PMID 18432533
- [Background] Yeung CK, Sihoe JD, Sit FK, Bower W, Sreedhar B, Lau J. Characteristics of primary nocturnal enuresis in adults: an epidemiological study. BJU Int. 2004 Feb;93(3):341-5. doi: 10.1111/j.1464-410x.2003.04612.x. PMID 14764133
- [Background] Van Tijen NM, Messer AP, Namdar Z. Perceived stress of nocturnal enuresis in childhood. Br J Urol. 1998 May;81 Suppl 3:98-9. doi: 10.1046/j.1464-410x.1998.00018.x. No abstract available. PMID 9634030
- [Background] Hagglof B, Andren O, Bergstrom E, Marklund L, Wendelius M. Self-esteem in children with nocturnal enuresis and urinary incontinence: improvement of self-esteem after treatment. Eur Urol. 1998;33 Suppl 3:16-9. doi: 10.1159/000052236. PMID 9599731
- [Background] Neveus T, Eggert P, Evans J, Macedo A, Rittig S, Tekgul S, Vande Walle J, Yeung CK, Robson L; International Children's Continence Society. Evaluation of and treatment for monosymptomatic enuresis: a standardization document from the International Children's Continence Society. J Urol. 2010 Feb;183(2):441-7. doi: 10.1016/j.juro.2009.10.043. Epub 2009 Dec 14. PMID 20006865
- [Background] Yeung CK, Chiu HN, Sit FK. Bladder dysfunction in children with refractory monosymptomatic primary nocturnal enuresis. J Urol. 1999 Sep;162(3 Pt 2):1049-54; discussion 1054-5. doi: 10.1016/S0022-5347(01)68062-5. PMID 10458430
- [Background] Hunsballe JM, Hansen TK, Rittig S, Pedersen EB, Djurhuus JC. The efficacy of DDAVP is related to the circadian rhythm of urine output in patients with persisting nocturnal enuresis. Clin Endocrinol (Oxf). 1998 Dec;49(6):793-801. doi: 10.1046/j.1365-2265.1998.00587.x. PMID 10209568
- [Background] Rittig S, Knudsen UB, Norgaard JP, Pedersen EB, Djurhuus JC. Abnormal diurnal rhythm of plasma vasopressin and urinary output in patients with enuresis. Am J Physiol. 1989 Apr;256(4 Pt 2):F664-71. doi: 10.1152/ajprenal.1989.256.4.F664. PMID 2705537
- [Background] Neveus T, Lackgren G, Tuvemo T, Hetta J, Hjalmas K, Stenberg A. Enuresis--background and treatment. Scand J Urol Nephrol Suppl. 2000;(206):1-44. PMID 11196246
- [Background] Kamperis K, Hagstroem S, Rittig S, Djurhuus JC. Combination of the enuresis alarm and desmopressin: second line treatment for nocturnal enuresis. J Urol. 2008 Mar;179(3):1128-31. doi: 10.1016/j.juro.2007.10.088. Epub 2008 Jan 18. PMID 18206924
- [Background] Dodds PR. Re: Evaluation of and treatment for monosymptomatic enuresis: a standardization document from the International Children's Continence Society: T. Neveus, P. Eggert, J. Evans, A. Macedo, S. Rittig, S. Tekgul, J. Vande Walle, C. K. Yeung and L. Robson J Urol 2010; 183: 441-447. J Urol. 2010 Aug;184(2):806-7; author reply 807-8. doi: 10.1016/j.juro.2010.04.006. No abstract available. PMID 20579671
- [Background] Andersen RF, Palmfeldt J, Jespersen B, Gregersen N, Rittig S. Plasma and urine proteomic profiles in childhood idiopathic nephrotic syndrome. Proteomics Clin Appl. 2012 Aug;6(7-8):382-93. doi: 10.1002/prca.201100081. PMID 22927352
- [Background] Rittig S, Frokiaer J. Basis and therapeutical rationale of the urinary concentrating mechanism. Int J Clin Pract Suppl. 2007 Sep;(155):2-7. doi: 10.1111/j.1742-1241.2007.01461.x. PMID 17727573
- [Background] Fernandez-Guerra P, Birkler RI, Merinero B, Ugarte M, Gregersen N, Rodriguez-Pombo P, Bross P, Palmfeldt J. Selected reaction monitoring as an effective method for reliable quantification of disease-associated proteins in maple syrup urine disease. Mol Genet Genomic Med. 2014 Sep;2(5):383-92. doi: 10.1002/mgg3.88. Epub 2014 Jun 4. PMID 25333063